CLINICAL TRIAL: NCT00981565
Title: Operative Versus Conservative Treatment in Mild Carpal Tunnel Syndrome, Randomized Prospective Multicenter Study
Brief Title: Mild Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, MD, North Karelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKCH-Surg-005
Record Dates: First submitted 2009-09-11; First posted 2009-09-22 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; CTS; medianus impingement
MeSH Terms: conditions — Carpal Tunnel Syndrome

ARMS (2):
- Operative (Active Comparator)
  Interventions: Procedure: open carpal tunnel release
- Conservative (Active Comparator)
  Interventions: Other: Night-cast

INTERVENTIONS:
Procedure: open carpal tunnel release — surgery to release the carpal tunnel
  Arms: Operative
Other: Night-cast — individual night time splinting
  Arms: Conservative

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral nerve entrapment. Diagnosis is based on symptoms, clinical findings and electrophysiological examination. Several conservative and surgical treatment options have been described.

Studies of surgical versus conservative treatment in mild carpal tunnel syndrome have not been done and it is still unclear whether or not surgical treatment is better than conservative treatment.

The aim of this study is to research has surgery better outcome in mild CTS than conservative treatment. Patient satisfactory, clinical and electrophysiologic outcomes, direct and indirect costs will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* electrophysiologically proven minimal or mild CTS lasting more than six months will be included in this study

Exclusion Criteria:

* rheumatoid arthritis
* diabetes mellitus
* hypothyreosis
* pregnancy
* wrist trauma or previous surgery
* splinting or corticosteroid injection on the affected side

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity Score | 1 year
Pain Visual Analogue Scale (VAS) | 1 year

SECONDARY OUTCOMES:
Change in electroneuromyography | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Finland (3):
  - North-Carelia Central Hospital, Joensuu
  - Kuopio University Hospital, Kuopio
  - Central Hospital of Mikkeli, Mikkeli